CLINICAL TRIAL: NCT02806804
Title: Safety and Immunogenicity Study of Quadrivalent Influenza Virus Vaccine in Healthy People Aged Years 3-60
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: cycdc2016-1
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Quadrivalent Influenza Virus Vaccine
Keywords: vaccine; safety; immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- one dose test vaccine (Experimental): One dose of quadrivalent influenza virus vaccine will be randomly given in aged 3-60 years old.
  Interventions: Biological: one dose test vaccine
- one dose commercially available trivalent influenza vaccine (Experimental): One dose of trivalent influenza virus vaccine will be randomly given in aged 3-60 years old.
  Interventions: Biological: one dose commercially available trivalent influenza vaccine
- One dose quadrivalent influenza virus vaccine (Experimental): One dose of quadrivalent influenza virus vaccine (trivalent influenza virus vaccine added to a new influenza B component) will be randomly given in aged 3-60 years old.
  Interventions: Biological: One dose of Quadrivalent Influenza Virus Vaccine

INTERVENTIONS:
Biological: one dose test vaccine
  Arms: one dose test vaccine
Biological: one dose commercially available trivalent influenza vaccine
  Arms: one dose commercially available trivalent influenza vaccine
Biological: One dose of Quadrivalent Influenza Virus Vaccine
  Arms: One dose quadrivalent influenza virus vaccine

SUMMARY:
This study evaluates the safety and immunogenicity of the quadrivalent influenza virus vaccine in healthy people aged years 3-60.Subjects will be randomly divided into 3 groups,receiving the test vaccine, commercially available trivalent influenza vaccine and trivalent influenza vaccine containing new influenza B component respectively. Each group has 800 subjects,2400 in total.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects more than 3 years old, and the subjects can be informed consent, and sign the informed consent.
* the subjects and his guardians can obey the demands of the scheme .
* Axillary temperature less than 37℃

Exclusion Criteria:

* The people who has flu or influenza-like symptoms(fever <axillary temperature ≥38 ℃>, cough or sore throat) within 3 months
* The people who has vaccinated influenza vaccine in 3years.
* The people who has a vaccine allergies, or who allergic to any kind of composition in experimental vaccine, such as eggs, ovalbumin etc.
* The people who has serious side effects to vaccine, such as allergy, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain.
* the subject who has symptoms of acute infection within a week.
* Autoimmune diseases or Immune function defect, people has immunosuppressive therapy, cytotoxic treatment or inhaled corticosteroids in the past 6 months.
* People has congenital malformations, developmental disorder or serious chronic diseases( such as Down's syndrome, diabetes, Sickle cell anemia or nerve system disease)
* People has asthma Unstable that need emergency treatment, hospitalization, intubation, oral or intravenous corticosteroid in the past 2 years.
* Diagnosed abnormal coagulation(Lack of clotting factors,Clotting disorders,Platelet abnormality) or significant bruising or coagulopathy
* people has history or family history of convulsions, seizures, encephalopathy and psychiatric.
* alienia, functional asplenia, and alienia or splenectomy in any situation.
* Serious neurological disorders such as Green Barry syndrome.
* people who has received blood products or immunoglobulin products in the past one months.
* people who has received other study drug in the past one month.
* people who received live attenuated vaccine, subunit vaccine or inactivated vaccine.
* people who has received allergy treatment in in the past 14 days.
* People who is on anti-TB treatment.
* People whose axillary temperature is more than 37℃ before the vaccination.
* People who is pregnant.
* Any factors unsuitable for clinical trail according to the researchers.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2400 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Evaluate serum antibody titers of quadrivalent influenza Vaccine in healthy people. | 28 days
  The serum antibody titers will be evaluated at 28 days after vaccination.
Evaluate the Rate of Adverse reactions of quadrivalent influenza Vaccine in healthy people. | 28 days
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy.